CLINICAL TRIAL: NCT00562029
Title: Modified Duodenal Switch Procedure "Duodenal-Jejunal Bypass" (Diabetes Surgery) As A Potential Cure for Type 2 Diabetes Mellitus in Non-Obese Patients- a Pilot Project to Validate a Prospective Randomized Control Trial
Brief Title: Study of Duodenal-Jejunal Bypass(DJB) as a Potential Cure for Type 2 Diabetes Mellitus
Acronym: DJB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sound Shore Medical Center of Westchester (Other)
Collaborators: Maffucci L, Rangraj M (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: djb-2007
Record Dates: First submitted 2007-11-19; First posted 2007-11-21 (Estimated); Last update posted 2015-05-21 (Estimated); Status verified 2015-05

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Diabetes Mellitus; Surgery; Duodenal Bypass; Resolution; Surgical Procedures
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- DJB patient (Experimental): Patient has undergone a duodeno-jejunal bypass
  Interventions: Procedure: Duodenal-jejunal Bypass

INTERVENTIONS:
Procedure: Duodenal-jejunal Bypass — Patient has undergone a duodenal bypass and bypass of 60cm of proximal jejunum

SUMMARY:
Premise: Complete resolution of Type 2 Diabetes Mellitus with normalization of blood glucose and HbA1c in the abscence of medication support is possible with a surgical procedure named the "Duodenal-Jejunal Bypass (DJB)" a modification of an established duodenal switch procedure and is performed utilizing the laparoscopic approach.

DETAILED DESCRIPTION:
Hypothesis: The duodenum plays a major role in glucose homeostasis through mechanisms largely unknown at this time. Evidence of this hypothesis comes from accumulated data in bariatric surgery patients who underwent Roux-en-y Gastric Bypass or Biliopancreatic Diversion (BPD) with or without a Duodenal Switch. Current evidence strongly supports this hypothesis with a long term (over 10 years) Type 2 Diabetes Mellitus(T2DM) resolution rate of 84-86% following the gastric bypass and over 95% for the duodenal switch.

The clinical resolution of T2DM is defined as independence of all anti-diabetic medications and maintaining a HbA1c less than 6.0. Recent rodent experiments by Francesco Rubino and subsequent human case reports by Cohen et al. supports the validity of this hypothesis. The modified procedure involved a roux-en-y bypass of the duodenum and 30-50cm of proximal jejunum, unaltering the stomach and pylorus resulted in resolution of T2DM with no weight loss in all subjects.

ELIGIBILITY:
Inclusion Criteria:

* Established diagnosis of Type 2 diabetes mellitus
* Body Mass Index(BMI) less than 35
* Insulin usage duration less than 10 years
* Negative anti-GAD
* Fasting C-peptide level over 1.0 mcg/ml
* Ability and willingness to follow up for a period of 1 year
* Willingness to consent for utilizing personal results without individual identifier information to be published in medical studies and other media as determined by the study investigators
* Ability to understand and describe the risks, benefits and mechanism of action of the procedure

Exclusion Criteria:

* Current pregnancy or positive pregnancy test
* Liver Cirrhosis
* Coagulopathy
* Type 1 Diabetes Mellitus
* HIV
* Previous abdominal surgery preventing laparoscopy
* Previous vagotomy
* Previous gastric or small intestine surgery
* Inability to comply with study requirements
* Currently active medical malpractice lawsuit/s
* Diseases of the exocrine pancreas: pancreatitis trauma, pancreatectomy, neoplasia, cystic fibrosis, hemochromatosis
* Endocrinopathies: acromegaly, glucagonoma, Cushing's Syndrome, pheochromocytoma, hyperthyroidism, somatostatinoma, aldorestanoma
* Chemical Induced Diabetes: vacor, pentamidine, nicotinic acid, glucocorticoids, thyroid hormones, diazoxide, beta-adrenergic agonists, thiazides, phenytoin, alfa-interferon
* Genetic Syndromes with Diabetes: Down's, Klinefelter's, Turner's, Wolfram, Lawrence-Moon- Beidel, Prader-Willi, Friederich's ataxia, Huntington's Chorea, Myotonic Dystrophy, Porphyria,
* If a candidate is deemed to be not an appropriate candidate based on investigators recommendation.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2007-11; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Measure: Resolution of Type 2 Diabetes Mellitus | One year

SECONDARY OUTCOMES:
Measure: Safety and efficacy of duodenal-jejunal bypass | One year

CONTACTS AND LOCATIONS:
Overall Officials: Leonard Maffucci, MD, Principal Investigator — Sound Shore Medical Center of Westchester; Madhu S Rangraj, MD, Principal Investigator — Sound Shore Medical Center of Westchester
Locations (1):
- Sound Shore Medical Center of Westchester, New Rochelle, New York, United States

REFERENCES:
- [Background] Rubino F, Forgione A, Cummings DE, Vix M, Gnuli D, Mingrone G, Castagneto M, Marescaux J. The mechanism of diabetes control after gastrointestinal bypass surgery reveals a role of the proximal small intestine in the pathophysiology of type 2 diabetes. Ann Surg. 2006 Nov;244(5):741-9. doi: 10.1097/01.sla.0000224726.61448.1b. PMID 17060767
- [Background] Buchwald H, Avidor Y, Braunwald E, Jensen MD, Pories W, Fahrbach K, Schoelles K. Bariatric surgery: a systematic review and meta-analysis. JAMA. 2004 Oct 13;292(14):1724-37. doi: 10.1001/jama.292.14.1724. PMID 15479938
- [Result] Cummings DE, Overduin J, Foster-Schubert KE, Carlson MJ. Role of the bypassed proximal intestine in the anti-diabetic effects of bariatric surgery. Surg Obes Relat Dis. 2007 Mar-Apr;3(2):109-15. doi: 10.1016/j.soard.2007.02.003. No abstract available. PMID 17386391
- [Result] Cohen RV, Schiavon CA, Pinheiro JS, Correa JL, Rubino F. Duodenal-jejunal bypass for the treatment of type 2 diabetes in patients with body mass index of 22-34 kg/m2: a report of 2 cases. Surg Obes Relat Dis. 2007 Mar-Apr;3(2):195-7. doi: 10.1016/j.soard.2007.01.009. No abstract available. PMID 17386401
- See also: click here for information on background to present study — http://ees.elsevier.com/soard/